CLINICAL TRIAL: NCT04420039
Title: Is Useful a Coaxial Plastic Stent Within a Lumen-Apposing Metal Stent For The Palliative Management Of Malignant Biliary Obstruction?
Brief Title: Plastic Stent Within a Lumen-Apposing Stent for Malignant Biliary Obstruction
Acronym: LAMSpigBil
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Joan B Gornals, Programme Director, Endoscopy Area, MD, PhD, Hospital Universitari de Bellvitge
Other Study IDs: HUBellvitge
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Cancer; Endoscopy; Oncologic Disorders; Therapy Related Neoplasms
Keywords: Malignant biliary obstrucction; Therapeutic endoscopy; Biliary drainage; Lumen apposing stent; Endoscopic Ultrasound; Pancreatic neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms, Second Primary | interventions — Choledochostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- 1- Single biliary LAMS: Unresectable/inoperable biliopancreatic cases with distal biliary obstruction who underwent EUS-BD with a single lumen-apposing stent after failed ERCP cannulation or inaccessible papilla.
  Interventions: Device: Endoscopic biliary transmural drainage
- 2- Biliary LAMS plus Doublu-Pigtail plastic Etent: Unresectable/inoperable biliopancreatic cases with distal biliary obstruction who underwent EUS-BD with a single lumen-apposing stent (plus double-pigtail plastic stent) after failed ERCP cannulation or inaccessible papilla.
  Interventions: Device: Endoscopic biliary transmural drainage

INTERVENTIONS:
Device: Endoscopic biliary transmural drainage — Endosonography-guided biliodigestive anastomosis using a dedicated biliary lumen-apposing stent in order to proveide a biliary drainage in cases of palliative malignant biliary obstruction.
  Two different strategies will be compared: single lumen-apposing stent vs lumen-apposing stent plus dousble-pigtail plastic stent.
  Other Names: Endoscopic Ultrasound-guided biliary drainage; Choledochoduodenostomy

SUMMARY:
There are doubts concerning the possible benefits derived from the insertion of double-pigtail plastic stents (DPS) within the lumen-apposing metal stents (LAMS) in the EUS-guided transmural biliary drainage (BD). The aims was to evaluate the safety of LAMS with and without a coaxial DPS in EUS-BD for the palliative management in malignant biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive unresectable/inoperable biliopancreatic cases with distal biliary obstruction who underwent EUS-BD after failed ERCP cannulation or inaccessible papilla

Exclusion Criteria:

* Borderline cancer cases
* Others type of biliary stents
* Severe coagulopathy or thrombocytopenia.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Palliative malignant biliopancreatic pathology
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Potential benefits | 4 weeks
  to respond if a coaxial DPS within a biliary LAMS really has a potential benefit in the EUS-BD (less number of adverse events: cholangitis, bleeding, sump syndrome, cholestasis secondary to stent biliary obstruction)

SECONDARY OUTCOMES:
Technical success | 24 hours
  Technical success was defined as a successful stent placement between the extrahepatic bile duct and duodenal lumen in a single step approach and determined by endoscopy and fluoroscopy
Clinical success | 4 weeks
  Clinical success was defined as a reduction in bilirubin by 50% at 2-weeks after stent placement, meaning that the biliary stent was functional.
Procedure time | 2 hours
  Procedure time was defined from the insertion of the endoscope to its removal.
Biliary reintervention | 6 months
  Biliary reintervention: the need to perform additional interventions to achieve biliary drainage.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Sant Pau i de la Santa Creu, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No